CLINICAL TRIAL: NCT00285350
Title: A Trial of Mycophenolate Mofetil in Myasthenia Gravis
Brief Title: Mycophenolate Mofetil in Myasthenia Gravis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: FDA Office of Orphan Products Development (U.S. Federal Agency)
Collaborators: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2154; NCT00127894 (obsolete NCT alias)
Record Dates: First submitted 2006-01-31; First posted 2006-02-02 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2007-03

CONDITIONS: Myasthenia Gravis
Keywords: myasthenia gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: mycophenolate mofetil

SUMMARY:
This is a prospective, multi-center, double-blind, placebo-controlled trial to determine the efficacy and safety of mycophenolate mofetil (MM) in combination with prednisone as the initial form of immunosuppression in patients with acquired myasthenia gravis (MG).

DETAILED DESCRIPTION:
80 patients with seropositive MG at 18 academic centers will be randomized to 3 months of treatment with 2.5 gm MM/day (1,250 mg q 12 hours, +/- 2 hours) plus 20 mg prednisone/day versus placebo plus 20 mg/day prednisone. The primary measure of efficacy will be the change from baseline in Quantitative MG (QMG) score at the end of 3 months. Secondary outcome measures include survival analysis for treatment failure, MG-related impairment of daily activities, functional assessment, manual muscle testing, SF-36 Health Status, and serum concentration of antibodies to the acetylcholine receptor. Study completers will have the option of taking open-label MM for an additional 6 months, during which prednisone will be reduced to the lowest dose necessary to maintain the optimum clinical response.

ELIGIBILITY:
Inclusion criteria

1. Acquired generalized MG diagnosed by one of the Principal Investigators based on:

   * Examination by site PI showing myasthenic weakness that is not limited to the ocular or peri-ocular muscles.
   * Elevated acetylcholine receptor antibodies.
   * Positive edrophonium chloride test or abnormal neuromuscular transmission demonstrated by single fiber EMG or repetitive nerve stimulation.
2. Aged at least 18.
3. Able to give informed consent.
4. Taking a constant dose of Mestinon for at least 2 weeks.
5. Symptom severity that would, in the judgment of the site investigator, justify initiation of immunosuppressive treatment.
6. Able and willing to comply with study requirements.

Exclusion criteria

1. Thymoma now or in the past.
2. Plasma exchange or IVIG treatment within 90 days of randomization.
3. Treatment with azathioprine, cyclosporine, mycophenolate mofetil, or other immunosuppressive medication since onset of MG. Treatment with prednisone or other corticosteroids within the previous 90 days.

   • Exception: patients may have taken doses of these immunosuppressant medications that are judged by the Principal Investigator to have been clinically insignificant, i.e. unlikely to produce improvement in MG.
4. Women of childbearing potential who are pregnant, breast-feeding or not practicing effective contraception.
5. Renal failure, active thyroid or hepatocellular disease, chronic infection, poorly controlled cardiac disease, or any other illness, including psychiatric disease, that would, in the opinion of the treating physician, make it unsafe for the patient to participate or would interfere with the interpretation of study results.
6. Weakness affecting only ocular or peri-ocular muscles (Myasthenia Gravis Foundation of America Class I).
7. Severe weakness predominantly affecting oropharyngeal, respiratory muscles or both (MGFA Class IVB).
8. Crisis or impending crisis (defined as FVC <10ml/Kg or bulbar weakness severe enough to compromise airway protection.)
9. Hemoglobin <10mg/dl; WBC <3,500.
10. History of non-compliance with treatment and office visits.
11. Thymectomy within 12 months before randomization.
12. Concurrent medical condition that would pose an unacceptable risk from immunosuppression, including a positive skin test for tuberculosis (PPD), unless the patient has previously received appropriate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80
Dates: Start 2002-09; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
QMGS

SECONDARY OUTCOMES:
Multiple

CONTACTS AND LOCATIONS:
Overall Officials: Donald B Sanders, MD, Principal Investigator — Duke University